CLINICAL TRIAL: NCT02860507
Title: A Randomized, Blinded-assessor, Single Center Study to Determine if Administration of Sugammadex, When Used to Reverse Deep Neuromuscular Blockade (NMB) After Open Abdominal Surgery, Impacts Hospital Efficiency
Brief Title: Study to Determine if Administration of Sugammadex Impacts Hospital Efficiency
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Enrico Camporesi, Attending Anesthesiologist & Director of Research, SE, University of South Florida
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TGH015
Record Dates: First submitted 2016-08-02; First posted 2016-08-09 (Estimated); Results first posted 2019-04-12 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Neuromuscular Blockade
MeSH Terms: interventions — Sugammadex; Neostigmine; Glycopyrrolate

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Double Blinded
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, Care Providers, Investigators, and Outcome Assessors are blinded from the type of NMBA reversal agent used prior to completion of data collection
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neostigmine + Glycopyrrolate (Active Comparator): Neostigmine 0.06 mg/kg and Glycopyrrolate 0.04mg/kg iv
  Interventions: Drug: Neostigmine; Drug: Glycopyrrolate
- sugammadex (Experimental): Sugammadex 4mg/kg
  Interventions: Drug: sugammadex

INTERVENTIONS:
Drug: sugammadex
  Other Names: Bridion
  Arms: sugammadex
Drug: Neostigmine
  Arms: Neostigmine + Glycopyrrolate
Drug: Glycopyrrolate
  Arms: Neostigmine + Glycopyrrolate

SUMMARY:
The purpose of this study is to evaluate the efficacy of Sugammadex in rapidly reversing deep neuromuscular blockaded (induced by rocuronium)

DETAILED DESCRIPTION:
Participants in the study group will receive a single bolus of Sugammadex (4.0mg/kg) prior to extubation. In the post-anesthesia care unit (PACU), a blinded safety-assessor will use the visual analog scale to clinically assess post-operative pain. Post-operative nausea and vomiting (PONV) will be assessed using a PONV rating scale every 30 minutes until PACU discharge. All patients will be monitored with continuous pulse-oximetry.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for open ventral hernia repair or open colectomy
* ASA class I-III
* 18 years and older
* Subjects with a body mass index (BMI) of <45kg/m2 and weight less than 150kg
* Subjects who have given written informed consent

Exclusion Criteria:

* Subjects with medical conditions and/or undergoing surgical procedures that are not compatible with the use of the TOF-Watch® SX (e.g., injuries to the thumbs/distal forearms, bilateral ulnar nerve damage or subjects with cardiac pacemaker
* Subjects known or suspected to have neuromuscular disorders impairing neuromuscular blockade (e.g., subjects with myasthenia gravis)
* Subjects known or suspected to have significant renal dysfunction (e.g. creatinine clearance < 30 mL.min-1
* Subjects known or suspected to have a (family)history of malignant hyperthermia; have significant hepatic dysfunction
* Subjects known or suspected to have an allergy to opiates/opioids, muscle relaxants or other medications used during general anesthesia;
* Subjects known or suspected to be hypersensitive to Sugammadex or other cyclodextrins or Rocuronium or any of its excipients
* Subjects who have a contraindication to, Rocuronium or Sugammadex
* Female subjects who are pregnant
* Morbidly obese subjects with a BMI > 45 kg/m2 or weight more than 150 kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Turner DA, Smith G. Evaluation of the combined effects of atropine and neostigmine on the lower oesophageal sphincter. Br J Anaesth. 1985 Oct;57(10):956-9. doi: 10.1093/bja/57.10.956. PMID 4041322
- [Background] Proakis AG, Harris GB. Comparative penetration of glycopyrrolate and atropine across the blood--brain and placental barriers in anesthetized dogs. Anesthesiology. 1978 May;48(5):339-44. doi: 10.1097/00000542-197805000-00007. No abstract available. PMID 646152
- [Background] Chhibber AK, Lustik SJ, Thakur R, Francisco DR, Fickling KB. Effects of anticholinergics on postoperative vomiting, recovery, and hospital stay in children undergoing tonsillectomy with or without adenoidectomy. Anesthesiology. 1999 Mar;90(3):697-700. doi: 10.1097/00000542-199903000-00010. PMID 10078669
- [Background] Tramer MR, Fuchs-Buder T. Omitting antagonism of neuromuscular block: effect on postoperative nausea and vomiting and risk of residual paralysis. A systematic review. Br J Anaesth. 1999 Mar;82(3):379-86. doi: 10.1093/bja/82.3.379. PMID 10434820
- [Background] Cheng CR, Sessler DI, Apfel CC. Does neostigmine administration produce a clinically important increase in postoperative nausea and vomiting? Anesth Analg. 2005 Nov;101(5):1349-1355. doi: 10.1213/01.ANE.0000180992.76743.C9. PMID 16243993
- [Background] Naguib M, Brull SJ. Update on neuromuscular pharmacology. Curr Opin Anaesthesiol. 2009 Aug;22(4):483-90. doi: 10.1097/ACO.0b013e32832b8cff. PMID 19384229
- [Background] Puhringer FK, Rex C, Sielenkamper AW, Claudius C, Larsen PB, Prins ME, Eikermann M, Khuenl-Brady KS. Reversal of profound, high-dose rocuronium-induced neuromuscular blockade by sugammadex at two different time points: an international, multicenter, randomized, dose-finding, safety assessor-blinded, phase II trial. Anesthesiology. 2008 Aug;109(2):188-97. doi: 10.1097/ALN.0b013e31817f5bc7. PMID 18648227
- [Background] Plaud B, Meretoja O, Hofmockel R, Raft J, Stoddart PA, van Kuijk JH, Hermens Y, Mirakhur RK. Reversal of rocuronium-induced neuromuscular blockade with sugammadex in pediatric and adult surgical patients. Anesthesiology. 2009 Feb;110(2):284-94. doi: 10.1097/ALN.0b013e318194caaa. PMID 19194156
- [Background] Hemmerling TM, Zaouter C, Geldner G, Nauheimer D. Sugammadex--a short review and clinical recommendations for the cardiac anesthesiologist. Ann Card Anaesth. 2010 Sep-Dec;13(3):206-16. doi: 10.4103/0971-9784.69052. PMID 20826961
- [Background] Abad-Gurumeta A, Ripolles-Melchor J, Casans-Frances R, Espinosa A, Martinez-Hurtado E, Fernandez-Perez C, Ramirez JM, Lopez-Timoneda F, Calvo-Vecino JM; Evidence Anaesthesia Review Group. A systematic review of sugammadex vs neostigmine for reversal of neuromuscular blockade. Anaesthesia. 2015 Dec;70(12):1441-52. doi: 10.1111/anae.13277. PMID 26558858
- [Background] Koyuncu O, Turhanoglu S, Ozbakis Akkurt C, Karcioglu M, Ozkan M, Ozer C, Sessler DI, Turan A. Comparison of sugammadex and conventional reversal on postoperative nausea and vomiting: a randomized, blinded trial. J Clin Anesth. 2015 Feb;27(1):51-6. doi: 10.1016/j.jclinane.2014.08.010. Epub 2014 Dec 24. PMID 25544263
- [Background] Sasaki N, Meyer MJ, Malviya SA, Stanislaus AB, MacDonald T, Doran ME, Igumenshcheva A, Hoang AH, Eikermann M. Effects of neostigmine reversal of nondepolarizing neuromuscular blocking agents on postoperative respiratory outcomes: a prospective study. Anesthesiology. 2014 Nov;121(5):959-68. doi: 10.1097/ALN.0000000000000440. PMID 25225821
- [Background] Murphy GS, Szokol JW, Marymont JH, Greenberg SB, Avram MJ, Vender JS. Residual neuromuscular blockade and critical respiratory events in the postanesthesia care unit. Anesth Analg. 2008 Jul;107(1):130-7. doi: 10.1213/ane.0b013e31816d1268. PMID 18635478
- [Background] Herbstreit F, Peters J, Eikermann M. Impaired upper airway integrity by residual neuromuscular blockade: increased airway collapsibility and blunted genioglossus muscle activity in response to negative pharyngeal pressure. Anesthesiology. 2009 Jun;110(6):1253-60. doi: 10.1097/ALN.0b013e31819faa71. PMID 19417617
- [Background] Murphy GS, Szokol JW, Marymont JH, Greenberg SB, Avram MJ, Vender JS, Nisman M. Intraoperative acceleromyographic monitoring reduces the risk of residual neuromuscular blockade and adverse respiratory events in the postanesthesia care unit. Anesthesiology. 2008 Sep;109(3):389-98. doi: 10.1097/ALN.0b013e318182af3b. PMID 18719436
- [Background] Butterly A, Bittner EA, George E, Sandberg WS, Eikermann M, Schmidt U. Postoperative residual curarization from intermediate-acting neuromuscular blocking agents delays recovery room discharge. Br J Anaesth. 2010 Sep;105(3):304-9. doi: 10.1093/bja/aeq157. Epub 2010 Jun 24. PMID 20576632
- [Background] Della Rocca G, Pompei L, Pagan DE Paganis C, Tesoro S, Mendola C, Boninsegni P, Tempia A, Manstretta S, Zamidei L, Gratarola A, Murabito P, Fuggiano L, DI Marco P. Reversal of rocuronium induced neuromuscular block with sugammadex or neostigmine: a large observational study. Acta Anaesthesiol Scand. 2013 Oct;57(9):1138-45. doi: 10.1111/aas.12155. Epub 2013 Jul 14. PMID 23849107

RESULTS

PARTICIPANT FLOW:
Groups:
- Neostigmine + Glycopyrrolate: Neostigmine 0.06 mg/kg and Glycopyrrolate 0.04mg/kg iv
  Neostigmine
  Glycopyrrolate
- Sugammadex: Sugammadex 4mg/kg
  sugammadex
Period: Overall Study
Arm/Group | Neostigmine + Glycopyrrolate | Sugammadex
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Neostigmine + Glycopyrrolate | Sugammadex | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.3 (5.2) | 45.6 (6.4) | 45.2 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 14 | 13 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 10
  Not Hispanic or Latino | 21 | 19 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 18 | 22 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Operating Room (OR) Turnover Time When Using Sugammadex Instead of Combination of Neostigmine and Glycopyrrolate.
Time Frame: through start of next surgery, average of 2 hours
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Neostigmine + Glycopyrrolate | Sugammadex
Number analyzed (Participants) | 25 | 25
Minutes | 49.7 (16.18) | 49.45 (16.67)

2. Secondary Outcome: Number of Patients Who Experience Postoperative Nausea and Vomiting, Post-operative Pain, and Post-operative Complications
Time Frame: through discharge from hospital, average of 72 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Neostigmine + Glycopyrrolate | Sugammadex
Number analyzed (Participants) | 25 | 25
Participants | 8 | 10

ADVERSE EVENTS:
Time Frame: Two days: collecting informed consent, and surgery (3 hours).
Description: Study was purely observational, Interventions followed hospital standard of care practices
Arm/Group | Neostigmine + Glycopyrrolate | Sugammadex
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-09-22): https://cdn.clinicaltrials.gov/large-docs/07/NCT02860507/Prot_SAP_000.pdf
  • Informed Consent Form (2015-12-16): https://cdn.clinicaltrials.gov/large-docs/07/NCT02860507/ICF_001.pdf